CLINICAL TRIAL: NCT01422239
Title: A Smoking Cessation Treatment for Adult Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1007007059
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Nicotine Dependence
Keywords: smoking; treatment; perceived risks
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored behavioral counseling (Experimental): The focus of the first three sessions for participants receiving the tailored treatment will be their three most highly endorsed perceived risks of quitting. All participants will receive information about preparing for quit day in the second session and coping with withdrawal symptoms in the third session using the Mayo Clinic's "Smoke Free and Living It" manual. The last 5 counseling sessions will be based on perceived risks of quitting.
  Interventions: Behavioral: Tailored treatment
- Standard behavioral counseling (Active Comparator): The focus of the first three sessions for participants receiving the standard treatment will be the benefits of quitting smoking. All participants will receive information about preparing for quit day in the second session and coping with withdrawal symptoms in the third session using the Mayo Clinic's "Smoke Free and Living It" manual. All participants will receive identical counseling sessions during week 4-8 based on material from the Mayo Clinic manual.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Tailored treatment — 8 sessions of individual behavioral counseling. The first 3 sessions will be 45 minutes long and include 30 minutes tailored to the perceived risks of quitting most strongly held by each participant. The final 5 sessions will be 30 minutes long and include material from the Mayo Clinic's smoking cessation manual.
  Arms: Tailored behavioral counseling
Behavioral: Standard Treatment — 8 sessions of individual behavioral counseling. The first 3 sessions will be 45 minutes long and include 30 minutes focused on the benefits of quitting smoking. The final 5 sessions will be 30 minutes long and include material from the Mayo Clinic's smoking cessation manual.
  Arms: Standard behavioral counseling

SUMMARY:
The purpose of this study is to develop and pilot test a smoking cessation counseling that focuses on the perceived risks of quitting smoking (e.g., weight gain, managing cravings and negative affect, loss of enjoyment).

Aim 1: To develop the risk-based smoking cessation intervention.

Aim 2: To examine whether manualized smoking cessation counseling about the perceived risks of quitting is feasible to administer and acceptable to adult women who want to quit smoking.

Aim 3: To examine smoking cessation outcomes for women who receive the risk-based treatment in comparison to standard smoking counseling. It is expected that women who receive risk-based counseling will show better quit rates and a longer time to relapse than women who receive standard treatment.

DETAILED DESCRIPTION:
The purpose of this treatment development study is to design and pilot test a smoking cessation intervention in which counseling sessions are tailored to individual smokers' perceived risks of quitting. The feasibility, acceptability, and efficacy of the novel treatment will be examined through a pilot study in which female smokers will be randomly assigned to receive either the tailored treatment or a standard treatment. It is expected that participants receiving the tailored treatment will show higher rates of smoking abstinence than participants receiving the standard smoking cessation treatment at the end of the 8-week treatment and at one month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 64 years old
* Meet Diagnostic and Statistical Manual-IV (DSM-IV) criteria for nicotine dependence with Fagerström Test for Nicotine Dependence (FTND) score ≥4
* Smoke at least 15 cigarettes (3/4 pack) daily (averaged over 1 week, in the past 1 month) and have an expired breath carbon monoxide (CO) level ≥10
* At the time of initial evaluation, are motivated to quit smoking in the next 30 days.
* Have the capacity to give informed consent, and are English-speaking.

Exclusion Criteria:

* Have a positive urine drug screen or urine pregnancy test at baseline evaluation
* Meet DSM-IV criteria for alcohol or other drug abuse or dependence in the previous 6 months
* Meet DSM-IV criteria for a current diagnosis of major depressive disorder, panic disorder or post-traumatic stress disorder
* Meet DSM-IV criteria for a current or past diagnosis of bipolar disorder or schizophrenia
* Are currently receiving treatment for nicotine dependence (e.g., nicotine replacement therapy, bupropion, chantix)

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea H. Weinberger, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, Department of Psychiatry, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants began in August of 2011 an ended in September 2012. Recruitment methods included radio advertisements, ClinicalTrials.gov, Craig's List postings, flyers, and referrals from research colleagues in the Department of Psychiatry
Pre-assignment Details: 28 adults signed the consent form and 20 adults were randomized and began the study. The 8 participants who completed the consent procedures but were not randomized were either not eligible (drug use, n=3; psychiatric diagnoses, n=2; low smoking, n=1) or did not attend the first study appointment and did not respond to attempts to contact (n=2).
Groups:
- Tailored Behavioral Counseling: The focus of the first three sessions for participants receiving the tailored treatment will be their three most highly endorsed perceived risks of quitting. All participants will receive information about preparing for quit day in the second session, coping with withdrawal symptoms in the third session, and on coping with triggers and withdrawal in the forth session using the Mayo Clinic's smoking cessation manual. The focus of sessions 5-7 will be the three perceive risks of quitting that were not covered during the first three session (i.e., the three least highly endorsed risks). Session 8 will cover maintenance of smoking abstinence using the Mayo Clinic manual.
- Standard Behavioral Counseling: The focus of the first three sessions for participants receiving the standard treatment will be the benefits of quitting smoking. All participants will receive information about preparing for quit day in the second session and coping with withdrawal symptoms in the third session using the Mayo Clinic's smoking cessation manual. All of the material for sessions 4-8 for the standard behavioral counseling condition will cover topics from the Mayo Clinic's smoking cessation manual - Session 4: coping with triggers to smoke and nicotine withdrawal, Session 5: Stress Management, Session 6: Time Management and Self-Image, Session 7: Communication Skills and Wellness, Session 8: Focusing on the Future (maintenance of smoking abstinence).
Period: Overall Study
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling
Started | 14 | 6
Completed | 10 | 3
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8.4) | 45.8 (13.3) | 44.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Point-prevalence Smoking Abstinence Assessed at the End of the Trial and Measured by Self-report and Confirmed by Carbon Monoxide Levels
Description: point-prevalence smoking abstinence assessed at the end of the trial and measured by self-report (no smoking reported in the previous 7 days) and confirmed by carbon monoxide levels (CO levels < 5ppm)
Time Frame: Up to 8 weeks
Population: Participants who dropped out of the study were considered to be smoking.
Measure: Number; unit: participants
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling
Number analyzed (Participants) | 14 | 6
participants | 4 | 1

2. Secondary Outcome: Point-prevalence Smoking Abstinence Four Weeks After the End of the Trial Assessed by Self-report and Carbon Monoxide Levels
Description: point-prevalence smoking abstinence assessed at one month after the completion of counseling and measured by self-report (no smoking reported in the previous 7 days) and confirmed by carbon monoxide levels (CO levels < 5ppm)
Time Frame: 12 weeks
Population: participants who did not complete the appointment were considered to be smoking
Measure: Number; unit: participants
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling
Number analyzed (Participants) | 14 | 6
participants | 2 | 1

3. Secondary Outcome: Change in Smoking From Baseline to the Followup Assessment (Week 12)
Description: Change in number of cigarettes per day (CPD) (averaged over the previous week) from the baseline assessment (Week 0) to the followup assessment (Week 12) for participants who did not quit smoking during the study.
Time Frame: Week 0 (baseline), Week 12 (one month followup)
Population: Participants who completed the week 8 appointment and provided the number of cigarettes smoked per day were included.
Measure: Mean (Standard Deviation); unit: CPD
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling
Number analyzed (Participants) | 6 | 2
CPD | 4.4 (5.4) | 2.0 (1.5)

ADVERSE EVENTS:
Arm/Group | Tailored Behavioral Counseling | Standard Behavioral Counseling
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6

LIMITATIONS AND CAVEATS:
Small sample size, half to two-thirds of participants dropped out of the active study phase, half to one quarter did not complete the one month follow up. Female participants only results can not be generalized to men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes